CLINICAL TRIAL: NCT01158313
Title: Development and Validation of Clinician-administered Bedside Screening Method for Patients With Potential Swallowing Impairment
Brief Title: Bedside Screening Method for Patients With Potential Swallowing Impairment
Acronym: CABS
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: HCN-DYS
Record Dates: First submitted 2010-06-22; First posted 2010-07-08 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Deglutition Disorders; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thickener: Patients with history of swallowing difficulties associated with aging and/or neurological diseases including patients with:
  * neurodegenerative diseases.
  * non-progressive neurological diseases including stroke.
  * older patients including nursing home patients.
  Interventions: Dietary Supplement: Thickened supplement

INTERVENTIONS:
Dietary Supplement: Thickened supplement — New thickener to be mixed to liquid to obtain different viscosities such as nectar viscosity, honey viscosity, conservative spoon-thick viscosity (CST) and extreme spoon-thick viscosity (EST

SUMMARY:
Previous studies have shown that most patients with functional oropharyngeal dysphagia could be quickly, safely and accurately recognized by using a clinical bedside method developed by the investigative team as the volume-viscosity swallow test (V-VST) that systematically evaluates the main clinical signs and symptoms of safety and efficacy of swallowing and monitors pulse oximetry to improve the detection of patients with silent aspirations.The aim of this study is to validate this test for persons suspected of having swallowing impairment, using a new thickener, with respect to the Videofluoroscopy (VFS) method (treated as the gold standard).

ELIGIBILITY:
Inclusion Criteria:

* History of swallowing difficulties associated with aging and/or neurological diseases including patients with: -neurodegenerative diseases. -non-progressive neurological diseases including stroke. -older patients including nursing home patients.
* Age > 18 y
* Ability to give informed consent

Exclusion Criteria:

* Patients suffering idiosyncratic phenomena or who are allergic to any medication, especially iodinated contrast media
* Patients suffering major respiratory disease or undergoing any type of surgery in the three months prior to the study
* Patients with a background of alcohol dependence or other drug dependence
* Patient who cannot be expected to comply with treatment
* Patient currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 Patients suspected of having symptoms of swallowing impairment will be enrolled in the study as well as 14 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of oropharyngeal dysphagia. | 24 hour period
  Diagnostic accuracy in terms of sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of oropharyngeal dysphagia.
Sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of impairment of safety in swallowing. | 24 hour period
  Diagnostic accuracy in terms of sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of impairment of safety in swallowing.
Sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of impairment of efficacy in swallowing. | 24 hour period
  Diagnostic accuracy in terms of sensitivity and specificity of the V-VST relative to VFS using THICKENER, in the diagnosis of impairment of efficacy in swallowing.

SECONDARY OUTCOMES:
Sensitivities and specificities of the V-VST relative to VFS for individual signs of impaired safety and efficacy | 24 hour timeframe

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Mataro, Mataró, Spain

REFERENCES:
- [Derived] Rofes L, Arreola V, Mukherjee R, Swanson J, Clave P. The effects of a xanthan gum-based thickener on the swallowing function of patients with dysphagia. Aliment Pharmacol Ther. 2014 May;39(10):1169-79. doi: 10.1111/apt.12696. Epub 2014 Mar 13. PMID 24628492